CLINICAL TRIAL: NCT05866471
Title: Activating Neuroplasticity to ENHANCE the Perception Box Expanding Effects of Psilocybin
Brief Title: The ENHANCE Study: taVNS and Psilocybin
Acronym: ENHANCE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Tiny Blue Dot Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2024-0463; A538900 (Other: UW Madison); Protocol Version 12/30/25 (Other: UW Madison)
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Psychedelic Experiences; Vagus Nerve Stimulation
Keywords: Psilocybin; Psychedelics; Vagus Nerve Stimulation; Healthy Volunteer
MeSH Terms: interventions — Psilocybin; Psychiatric Rehabilitation

STUDY DESIGN:
Intervention Model Description: randomization will be stratified by sex
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Sham taVNS + Psilocybin + taVNS (Experimental): Group 1 will receive twice daily sham taVNS for 7 days immediately prior to psilocybin dosing. Post-psilocybin dosing, they will receive twice-daily taVNS paired with psychedelic session contextual cues for 7 days.
  Interventions: Drug: Psilocybin; Device: Transcutaneous auricular Vagus Nerve Stimulation (taVNS); Other: Sham taVNS
- Group 2: Sham taVNS + Psilocybin + Sham taVNS (Sham Comparator): Group 2 will receive twice daily sham taVNS for 7 days immediately prior to psilocybin dosing. Post-psilocybin dosing, they will receive twice-daily sham taVNS paired with psychedelic session contextual cues for 7 days.
  Interventions: Drug: Psilocybin; Other: Sham taVNS
- Group 3: Sham taVNS + Psilocybin + Psychosocial Support Alone (Active Comparator): Group 3 will receive twice daily sham taVNS for 7 days immediately prior to psilocybin dosing. Post-psilocybin dosing, they will receive psychosocial support alone, comprised of an integration session 1 day and 1-week post-psilocybin dosing. They will not receive active or sham taVNS post-psilocybin.
  Interventions: Drug: Psilocybin; Behavioral: Psychosocial Support Alone; Other: Sham taVNS
- Group 4: taVNS + Psilocybin + Sham taVNS (Active Comparator): Group 4 will receive twice daily taVNS for 7 days immediately prior to psilocybin dosing. Post-psilocybin dosing, they will receive twice-daily sham taVNS paired with psychedelic session contextual cues for 7 days.
  Interventions: Drug: Psilocybin; Device: Transcutaneous auricular Vagus Nerve Stimulation (taVNS); Other: Sham taVNS

INTERVENTIONS:
Drug: Psilocybin — The psilocybin is produced under Good Manufacturing Practice and is in a capsule that contains 25 mg of botanically-derived psilocybin.
  Other Names: Psilocybine, Psilocibin; Filament Health Psilocybin; PEX010
Device: Transcutaneous auricular Vagus Nerve Stimulation (taVNS) — For both the active and sham taVNS procedure, participants will be provided with, and trained on, taVNS devices that apply gentle stimulation to the left ear via either electrodes or an earpiece that fits over the left ear.
  Arms: Group 1: Sham taVNS + Psilocybin + taVNS; Group 4: taVNS + Psilocybin + Sham taVNS
Behavioral: Psychosocial Support Alone — Participants assigned to Psychosocial Support Alone will not receive taVNS following psilocybin dosing.
  Arms: Group 3: Sham taVNS + Psilocybin + Psychosocial Support Alone
Other: Sham taVNS — For both the active and sham taVNS procedure, participants will be provided with, and trained on, taVNS devices that apply gentle stimulation to the left ear via either electrodes or an earpiece that fits over the left ear.

SUMMARY:
This study will examine whether combining a single dose of psilocybin with non-invasive transcutaneous auricular vagus nerve stimulation (taVNS), a potential inducer of neuroplasticity and enhanced memory formation, will enhance the long-term beneficial behavioral effects of psilocybin when compared to sham taVNS or no VNS by allowing memory for insights gained during the psychedelic experience to remain vivid after they will have faded in subjects who receive psilocybin followed by sham taVNS or no VNS.

DETAILED DESCRIPTION:
One hundred and eight medically healthy adult volunteers with a modest decrement in wellbeing will receive a single open-label 25 mg dose of psilocybin administered within a "set and setting" (SaS) framework of psychological support provided by trained facilitators, such as has been successfully employed in prior psychedelic studies at UW-Madison. The SaS protocol will include 2-4 hours of preparation, a 6- to 8-hour psilocybin dosing session and an hour-long integration session 1 day and 9 days post dosing. All subjects will receive various combinations of active taVNS or sham taVNS prior to, or following, psilocybin dosing.

Active and sham taVNS sessions will last 20 minutes and will occur twice daily (morning and afternoon/evening) for 7 consecutive days, using an "at home" protocol that has been used safely and effectively by study collaborators. taVNS is a non-invasive low-risk procedure.

Subjects will be randomized with equal allocation to one of four conditions: 1) seven days of sham taVNS prior to psilocybin dosing and 7 days of active taVNS post- psilocybin dosing (Group 1: n=27); 2) seven days of sham taVNS prior to psilocybin dosing and 7 days of sham taVNS post- psilocybin dosing (Group 2: n=27); 3) seven days of sham taVNS prior to psilocybin dosing and psilocybin with psychosocial support post-dosing (Group 3: n=27); and 4) seven days of active taVNS prior to psilocybin dosing and 7 days of sham taVNS post- psilocybin dosing (Group 4: n=27). Importantly, participants in all groups will receive psychosocial support in addition to their randomization status (i.e., taVNS or sham taVNS prior to, or following psilocybin, or psychosocial support alone), as the provision of psychosocial support is the current standard of care for the use of psychedelics in FDA-regulated clinical trials (FDA 2023). It is anticipated that a total sample of 108 subjects will be enrolled to provide 100 subjects who complete study activities/assessments sufficient to provide evaluable data for testing study primary and exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Ability/willingness to complete all study activities
* Modest reduction in emotional well-being
* Medically healthy (does not meet criteria for an exclusionary medical condition)
* Blood pressure and heart rate within established ranges at screening
* Use of acceptable contraceptive methods (sexually active males and women of childbearing potential)

Exclusion Criteria:

* Clinically significant safety lab abnormalities (i.e., Complete Blood Count with Differential, Comprehensive Metabolic Panel, and urinalysis)
* Current or clinically significant psychiatric disorder that, in the investigator's judgment, would interfere with participation or increase risk
* Current use of drugs or medications, prescribed or otherwise, that may interact with psilocybin
* Use of investigational drugs, biologics, or devices within 30 days of enrollment
* Use of psychedelic or related agents within three months of Dosing Day
* Clinically significant electrocardiogram (ECG)
* Vitals outside acceptable range
* Pregnancy and currently breastfeeding
* Unwillingness to go without tobacco products for 12 hours or more
* Inability to undergo fMRI scanning
* Recent ear trauma, hearing loss (if clinically significant), or deafness
* Family history of a psychotic disorder in a first degree relative

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Memory Experiences Questionnaire (MEM-Q-PSIL): Comparison of taVNS Administration vs. Treatment as Usual | 8 weeks
  The MEM-Q is 31-item self-report scales designed to measure 10 phenomenological qualities of autobiographical memories: Vividness, Coherence, Accessibility, Time Perspective, Sensory Details, Visual Perspective, Emotional Intensity, Sharing, Distancing and Valence. Ratings are made on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
Functional Magnetic Resonance Imaging (fMRI): Comparison of taVNS Administration vs. Treatment as Usual | Day 1 and Day 56 Post- Psilocybin Dose
  Activation in brain regions associated with cued autobiographical memory retrieval will be assessed with fMRI. Group comparisons will examine differences in whole brain blood oxygenated level dependent (BOLD) signal and connectivity based on previously established seed-based methods using a priori brain regions implicated in autobiographical memory retrieval corresponding dosing session stimuli. The study team will update with more specific information when the details are confirmed.
Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS): Comparison of taVNS Administration vs. Treatment as Usual | 8 weeks
  The WEMWBS is a 14-item self-report scale that was designed to measure the psychological well-being of a population. The questions use a five-point Likert scale. The items are all worded positively and cover both feeling and functioning aspects of mental wellbeing. Items on the questionnaire are rated on a 5-point scale, where 1= "None of the time", 2= "rarely", 3= "some of the time", 4= "often", 5= "all the time". A total scale score is calculated by summing the 14 individual item scores. The total possible range of scores for the WEMWBS is 14-70 with higher scores indicating a greater well-being.
Summary of Adverse Events | up to 8 weeks
  Adverse events (AEs) categorized by CTCAE v5.0 criteria at all assessments (6 study visits).

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data including, but not limited to, demographics, questionnaires, adverse events, and fMRI data may be made available to qualified researchers upon request.
Time Frame: Following publication of primary study findings.
Access Criteria: All de-identified data will be made available to qualified researchers in a way that protects subject confidentiality and adheres to HIPAA policies. Both internal and external requests for data will be handled by the Principal Investigator (PI) to ensure equitable access, fairness, and safeguards. After reviewing a short proposal prepared by an external investigator, the PI will approve requests with appropriate experimental design, scientific merit, and Institutional Review Board (IRB) approval and recommend revisions for proposals requiring further justification or modifications. Informed consent documents will provide sufficient detail about the intent to archive, share, and re-analyze data.
  MRI data will also be shared upon request using the same data sharing process described above. To facilitate interpretation of the data, imaging parameters, gender, age, and racial information will be shared and associated with the dataset.